CLINICAL TRIAL: NCT03602716
Title: A Research on High-Definition Transcranial Direct Current Stimulation as a Treatment of Negative Symptoms in Patients With Schizophrenia
Brief Title: High-Definition Transcranial Direct Current Stimulation as a Treatment of Negative Symptoms of Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was recruited slowly due to the imapct of some uncontrollable factors, such as COVID19.
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17411970000
Record Dates: First submitted 2018-06-27; First posted 2018-07-27 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2020-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia; HD-tDCS; negative symptoms
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HD-tDCS group (Experimental): This HD-tDCS group will be stimulated by active HD-tDCS.
  Interventions: Device: HD-tDCS
- Sham HD-tDCS group (Sham Comparator): This sham HD-tDCS group will have a sham stimulation with HD-tDCS.
  Interventions: Device: Sham HD-tDCS

INTERVENTIONS:
Device: HD-tDCS — HD-tDCS is going to be delivered at 1.5 mA intensity for 20 minutes once a day (+15 s fade-in and fade-out); sessions will be performed on 10 days 5 consecutive weekdays with sustained effects at T1 and T2. HD-tDCS will be used with the anode placed over the left DLPFC (F3) surrounded by four cathodes at F5, F1, FC3, and AF3 based on the 10/20 international EEG system.
  Arms: HD-tDCS group
Device: Sham HD-tDCS — HD-tDCS is going to be used with the anode placed over the left DLPFC (F3) surrounded by four cathodes at F5, F1, FC3, and AF3 based on the 10/20 international EEG system; sessions will be performed on 10 days 5 consecutive weekdays with sustained effects at T1 and T2. This group will have a 20-min-sham stimulation.
  Arms: Sham HD-tDCS group

SUMMARY:
In this study, investigators designed a double-blind randomized trial to prove a more reliable evidence to show how the treatment by using high-definition transcranial direct current stimulation (HD-tDCS) can relieve negative symptoms in patients with predominant negative symptoms of schizophrenia, especially on improving participants' anhedonia condition and social cognition, through stimulating the left dorsolateral prefrontal cortex (DLPFC). Participants will be divided into active and sham HD-tDCS groups equally.

DETAILED DESCRIPTION:
Schizophrenia is one of the most disabling psychiatric disorders that almost 1% worldwide population suffer from this devastating illness. The clinical expression of this illness has been categorized into different dimensions, though most of the patients are well treated with antipsychotic medication, the negative symptom is still one of the very refractory symptoms. Emerging evidence shows that transcranial direct current stimulation (tDCS) is a promising treatment for schizophrenia negative symptoms, however, findings are still controversial. HD-tDCS can provide a more stable and accurate direct current comparing with traditional tDCS, which gives a hope to treat negative symptoms in a more reliable way.

An association between negative symptoms and grey matter reductions in the prefrontal cortex is found, moreover, even during rest, hypoactivity of the prefrontal cortex, particularly of the left dorsolateral, and of the anterior cingulate regions, has been linked to negative symptoms of schizophrenia. It has been observed that tDCS could relatively alleviate negative symptoms in patients with schizophrenia by stimulating the left DLPFC through an anodal electrode, which has been proved can also modulate brain functional connectivity and have clinical improvements.

Half of the participants with a clinical presentation of predominant negative symptoms will be stimulated by active HD-tDCS and the rest will have a sham stimulation. HD-tDCS is going to be delivered at 1.5 mA intensity for 20 minutes once a day; sessions will be performed on 10 days 5 consecutive weekdays with sustained effects at 1 (T2) and 3 (T3) months. A Soterix Medical 4x1 HD-tDCS will be used with the anode placed over the left DLPFC (F3), surrounded by four cathodal electrodes at F5, F1, FC3 and AF3, based on the 10/20 international EEG system. All the outcomes will be assessed at baseline (T0, before HD-tDCS sessions), one day after the 10th HD-tDCS sessions (T1), and also at T2 and T3. Both participants and investigators will be blind to this treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnostic schizophrenia by DSM-IV
* patients at an age between 18-60 years of Han nationality
* 1) baseline score equal or higher than 4 in at least two items in negative symptoms at PANSS; 2) or baseline score equal or higher than 3 points in at least 1/3 items (including apathy) for negative symptoms; and 3)No more than 2 items have a score higher than 3 points for positive symptoms at PANSS.
* willing to participate in the experiment and take treatment

Exclusion Criteria:

* other psychiatric diagnoses
* criteria for bipolar disorder; dementia; other psychotic disturbs; substance-related disorders
* schizophrenia caused by organic diseases
* other mental disorders caused by drugs and alcohol
* IQ<70
* presence of serious suicidal behaviour
* claustrophobic or pregnancy
* metal implantation in vivo
* specific tDCS limitations (such as anatomic problems and high sensitivity on current)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2020-09-26 (Actual)

PRIMARY OUTCOMES:
The Positive and Negative Syndrome Scale (PANSS) | Change from baseline through study completion and sustained effects at 1 and 3 months.
  a 30-items, 7-point rating scale; the 7 rating points represent increasing levels of psychopathology: 1= absent, 2= minimal, 3= mild, 4 = moderate, 5= moderate-severe, 6= severe, 7= extreme; of the 16 items, 7 were chosen to constitute Positive Scale, 7 items for Negative Scale and the remaining 16 items for a General Psychopathology Scale.
The Scale for the Assessment of Negative Symptoms (SANS) | Change from baseline through study completion and sustained effects at 1 and 3 months.
  a 24-items, 5-point rating scale; the 5 rating points represent increasing levels of psychopathology: 0= absent, 1= mild, 2= moderate, 3= severe, 4= extreme; of the 24 items, the first 6 items for Affective Flattening, 5 items for Alogia, 5 items for Avolition, 5 items for Anhedonia, and the remaining 3 items for Attention.
The Clinical Assessment Interview for Negative Symptoms (CAINS) | Change from baseline through study completion and sustained effects at 1 and 3 months.
  including CAINS and CAINS self-reported checklist

SECONDARY OUTCOMES:
the Temporal Experience of Pleasure Scale (TEPS) | Change from baseline through study completion and sustained effects at 1 and 3 months.
  a self-reported questionnaire
the Emotional Expression Scale (EES) | Change from baseline through study completion and sustained effects at 1 and 3 months.
  a self-reported questionnaire
the Belief About Pleasure Scales (BAPS) | Change from baseline through study completion and sustained effects at 1 and 3 months.
  a self-reported questionnaire
the Emotional Regulation Questionnaire (ERQ) | Change from baseline through study completion and sustained effects at 1 and 3 months.
  a self-reported questionnaire
the Beck Depression Inventory (BDI) | Change from baseline through study completion and sustained effects at 1 and 3 months.
  a self-reported questionnaire
the Effort Expenditure for Rewards Task (EEfRT) | Change from baseline through study completion and sustained effects at 1 and 3 months.
  a computer test
the Belief Updating Task | Change from baseline through study completion and sustained effects at 1 and 3 months.
  a computer test
the Anticipatory and Consummatory Pleasure (ACP) task performances | Change from baseline through study completion and sustained effects at 1 and 3 months.
  a computer test

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China